CLINICAL TRIAL: NCT06759077
Title: Potential Beneficial Cardio Protective Effect of SGL2I in Hemodialysis Patients and Its Impact on Patient Quality of Life
Brief Title: Cardio Protective Effect of SGL2I in Hemodialysis Patients and Its Impact on Patient Quality of Life
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, suzan.D.zakaria, Pharmacist at Clinical Pharmacy Department, Faculty of Pharmacy (Girls), Al-Azhar University Master Degree of Pharmaceutical Sciences (Clinical Pharmacy), Al-Azhar University (2023), Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: FWA 000017585
Record Dates: First submitted 2024-12-30; First posted 2025-01-06 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Kidney Diseases
MeSH Terms: conditions — Kidney Diseases | interventions — dapagliflozin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- standard treatment (No Intervention): Adult patients with advanced CKD who will take the standard treatment for 6months.
- interventional Group (Experimental): adult patients with advanced CKD who will take SGL2I(DAPAGLIFLOZINE at a dose (10 mg/day) orally for 6months
  Interventions: Drug: Dapagliflozin (DAPA)

INTERVENTIONS:
Drug: Dapagliflozin (DAPA) — adult patients with advanced CKD who will take SGL2I(DAPAGLIFLOZINE at a dose (10 mg/day) orally for 6months
  Arms: interventional Group

SUMMARY:
If this study has a cardio protective effect it will affect the mortality and morbidity of advanced CKD patients and improve their quality of life

DETAILED DESCRIPTION:
Cardiovascular disease is the leading cause of mortality, accounting for >50% of deaths with known causes, while cardiovascular mortality is 9-fold higher in these patients compared with age- and sex-matched individuals in the general population Particularly, heart failure poses a significant challenge in the management of ESKD. It frequently develops after initiation of dialysis and is a prominent mortality risk factor among these patients When CKD patients develop HF, increased sodium and fluid retention, and vascular tension will lead to increased preload of the heart. The increased ventricular wall pressure will lead to release biomarkers like natriuretic peptides (NP). Therefore, biomarkers of myocardial stretch are commonly used in the diagnosis and prognosis evaluation of HF. It is worth noting that the negative predictive value of NP is extremely high (0.94-0.98), while the positive predictive value is slightly lower, (0.44-0.57) for chronic heart failure (CHF) and (0.66-0.67) for acute heart failure (AHF), Commonly used myocardial stretch marker include NT-pro BNP .

NT-pro BNP has the advantage that Accuracy of negative diagnosis is extremely high; The prognostic value is the most powerful, especially in CKD stages 4-5 and dialysis patients Traditional therapies to prevent CVD complications in the general population have shown to be ineffective in Chronic kidney disease (CKD). To address the unmet need, further research is needed to evaluate novel therapeutic strategies to improve cardiovascular outcomes among patients on dialysis .

Over the last several years, Sodium-glucose transporter type 2 (SGLT2) inhibitors have been shown to confer substantial kidney and cardiovascular benefits among patients with type 2 diabetes, heart failure, and/or high-risk CKD .

Secondary analyses from these landmark trials demonstrated consistent benefits of SGLT2 inhibitors across many subgroups, supporting the widespread use and incorporation in clinical practice guidelines of this new kidney and cardio protective drug class.

ELIGIBILITY:
Inclusion Criteria:

* Patients with CKD stage5 (i.e., eGFR < 15 mL/min/1.73m2) (Inker et al., 2021)

Exclusion Criteria:

* patients who refuse to sign consent
* Patients with acute heart failure , will exclude patients with known prior ischemic heart diseases or ischemic cardiomyopathy
* Autosomal dominant polycystic kidney disease (ADPKD).
* Type 1 diabetes mellitus
* History of ketoacidosis in the last year.
* Known hypersensitivity to SGLT2 inhibitors.
* Known severe hepatic impairment (Child-Pugh class C)
* Pregnant or breastfeeding females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2024-12-28 (Actual); Primary Completion 2024-12-28 (Estimated); Study Completion 2025-12-28 (Estimated)

PRIMARY OUTCOMES:
Investigate the cardio protective effect of SGL2 inhibitors(DAPAGLIFLOZINE (10 mg/day)) in dialysis patients ,by measuring human N terminal pro brain natriuretic peptide (N -pro BNB) at baseline and after 6months | up to 24 weeks

SECONDARY OUTCOMES:
Assess the degree of quality of life by Heart Failure Patient Questionnaire to assess cardiac support in dialysis patients | up to 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of pharmacy (girls )ALAzhar university, Cairo, Egypt

REFERENCES:
- [Background] Kobo O, Abramov D, Davies S, Ahmed SB, Sun LY, Mieres JH, Parwani P, Siudak Z, Van Spall HGC, Mamas MA. CKD-Associated Cardiovascular Mortality in the United States: Temporal Trends From 1999 to 2020. Kidney Med. 2022 Dec 28;5(3):100597. doi: 10.1016/j.xkme.2022.100597. eCollection 2023 Mar. PMID 36814454
- [Background] Rashid AM, Jamil A, Khan Z, Shakoor M, Kamal UH, Khan II, Akram A, Shahabi M, Yamani N, Ali S, Fatima K, Kamdi A, Junaid M, Khan AM, Mattumpuram J, Perswani P. Trends in mortality related to kidney failure and diabetes mellitus in the United States: a 1999-2020 analysis. J Nephrol. 2024 Sep;37(7):1833-1841. doi: 10.1007/s40620-024-01990-z. Epub 2024 Jun 25. PMID 38916852
- [Background] McDonagh TA, Metra M, Adamo M, Gardner RS, Baumbach A, Bohm M, Burri H, Butler J, Celutkiene J, Chioncel O, Cleland JGF, Coats AJS, Crespo-Leiro MG, Farmakis D, Gilard M, Heymans S, Hoes AW, Jaarsma T, Jankowska EA, Lainscak M, Lam CSP, Lyon AR, McMurray JJV, Mebazaa A, Mindham R, Muneretto C, Francesco Piepoli M, Price S, Rosano GMC, Ruschitzka F, Kathrine Skibelund A; ESC Scientific Document Group. 2021 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure. Eur Heart J. 2021 Sep 21;42(36):3599-3726. doi: 10.1093/eurheartj/ehab368. No abstract available. PMID 34447992
- [Background] Han X, Zhang S, Chen Z, Adhikari BK, Zhang Y, Zhang J, Sun J, Wang Y. Cardiac biomarkers of heart failure in chronic kidney disease. Clin Chim Acta. 2020 Nov;510:298-310. doi: 10.1016/j.cca.2020.07.040. Epub 2020 Jul 23. PMID 32710942
- [Background] Siddiqui R, Obi Y, Dossabhoy NR, Shafi T. Is There a Role for SGLT2 Inhibitors in Patients with End-Stage Kidney Disease? Curr Hypertens Rep. 2024 Dec;26(12):463-474. doi: 10.1007/s11906-024-01314-3. Epub 2024 Jun 24. PMID 38913113
- [Background] McGuire DK, Shih WJ, Cosentino F, Charbonnel B, Cherney DZI, Dagogo-Jack S, Pratley R, Greenberg M, Wang S, Huyck S, Gantz I, Terra SG, Masiukiewicz U, Cannon CP. Association of SGLT2 Inhibitors With Cardiovascular and Kidney Outcomes in Patients With Type 2 Diabetes: A Meta-analysis. JAMA Cardiol. 2021 Feb 1;6(2):148-158. doi: 10.1001/jamacardio.2020.4511. PMID 33031522
- [Background] Kidney Disease: Improving Global Outcomes (KDIGO) Diabetes Work Group. KDIGO 2022 Clinical Practice Guideline for Diabetes Management in Chronic Kidney Disease. Kidney Int. 2022 Nov;102(5S):S1-S127. doi: 10.1016/j.kint.2022.06.008. No abstract available. PMID 36272764